CLINICAL TRIAL: NCT04011930
Title: Effects of Vitamin D3 Supplementation on Antioxidant Enzymes Level in Vitamin D3 Deficient COPD Patients
Brief Title: This Study Include Chronic Obstructive Pulmonary Disease(COPD) Patients . Patients Were Vitamin D Deficient Age Range 40 to 80 Years, Smokers Patients Were Advised to Take Either Placebo or Vitamin D3 . Antioxidant Enzymes Were Assessed at Baseline and at 26th Weeks.
Acronym: BSMMU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr Salma Anjum, MD RESIDENT, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7102
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol; Vitamin D; Calcitriol

STUDY DESIGN:
Intervention Model Description: All eligible patients were randomly assigned to either study (A) control(B) group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental study (Active Comparator): vitamin D Generic name -cholecalciferol (40,000IU)Dose-80,000 Dosage -2capsule/week for consecutive 26 weeks.
  Drug cholecalciferol- ingredients -cholecalciferol (40,000 IU) Microcrystalline cellulose(58.1 gm),hydroxy toluene (.2mg),magnesium stearate(3mg0,gelatin capsule shell(1mg)
  other name D-rise
  Interventions: Drug: cholecalciferol
- Experimental control (Placebo Comparator): Placebo oral capsule Dose-80,000 Dosage -2capsule/week for consecutive 26 weeks
  placebo oral capsule-ingredients-microcrystalline cellulose,butylated hydroxy toluene
  ,magnesium stearate
  other name D-rise
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: cholecalciferol — 80,000 IU(2 capsules)/week for 13 weeks and then according to the serum calcium and serum D level 40,000 IU/2 to 3 weeks for next 13 weeks
  Other Names: Vitamin D; Calcitriol
  Arms: Experimental study
Drug: Placebo oral capsule — 80,000 IU(2 capsules)/week for 13 weeks and then according to the serum calcium and serum D level 40,000 IU/2 to 3 weeks for next 13 weeks
  Other Names: placebo treatment
  Arms: Experimental control

SUMMARY:
Vitamin D3 supplementation dose not increase plasma antioxidant enzymes level in COPD patients was the null hypothesis of the research.

DETAILED DESCRIPTION:
On the first day of enrollment, the objectives, nature, purpose and potential risk of all the procedures which are intended to be used for the study will be explained in detail to each COPD patients (diagnosed by pulmonologist), with a cordial attitude giving emphasis on the benefits he might obtain from this study. He will be encouraged for voluntary participation and will be allowed to withdraw himself from the study even after participation, whenever he feels uneasy. If he will agree to be enrolled in the study, an informed written consent will be taken in a prescribed form. Details family history, medical history and thorough physical examination of each patient will be done and all the information will be recorded in a standard data sheet. Then all the patients will be requested to attend the Department of Physiology at 8:30 am (after overnight fasting) on the examination day.

On that day, 16 ml of venous blood will be collected from antecubital vein of patient in different vacutainer tubes and will be taken to the laboratory of Department of Biochemistry and Molecular Biology as soon as possible, where 3 ml will be used for the estimation of serum vitamin D3 and rest will be preserved at -4˚C.

If the patient is with serum 25(OH)D <30 ng/ml (D3 deficiency) but >10 ng/ml (severe D3 deficient; for ethical purpose), then the serum parathormone (PTH), serum calcium, serum inorganic phosphate, serum alkaline phosphatase (ALP), serum glutamate-pyruvate transaminase (SGPT), fasting blood glucose, serum glycosylated hemoglobin HbA1C, serum cholesterol, serum high density lipoprotein (HDL), serum low density lipoprotein (LDL), serum triglyceride (TG), serum creatinine will be assessed from the preserved blood. After getting all the biochemical reports the final selection will be done, according to the inclusion and exclusion criteria. In addition serum level of Catalase and Superoxide dismutase will be done in the Department of Physiology, BSMMU. Then all the eligible patients will be randomly assigned to either 'study (A)' or 'control (B)' group. These data will be recorded as values of 'day 0' (A0, B0).

Subsequently a standard therapeutic treatment (according to Global initiative for chronic obstructive pulmonary disease guideline) will be prescribed (by the pulmonologist) to all the selected stable COPD patients of both groups. Proper education will be given about drug, method of taking medication and medication plan.

Along with the standard pharmacological treatment of COPD, all patients of both the groups will be advised to have sunlight exposure (within 11 am to 2 pm) only for 20 minutes daily and also to continue ad lib (according to their own choice) diet. In addition, oral vitamin D3 (80,000 IU per week) and placebo will be added to the treatment schedule of the 'Study' patients and 'Control' patients, respectively, for consecutive 13 weeks.

Subsequently, all these patients (of both groups) will be cordially requested to attend the Department of Physiology on 13th week of their follow up, to reexamine the serum 25(OH)D and Calcium (to check the toxicity or deficiency). Then according to serum level of 25(OH)D and Ca, [vitamin D3 40,000 IU (1 capsule) per one to six weeks] (Vitamin D council 2019) will be again given to the 'Study' patients for further 13 weeks. On the other hand, if serum 25(OH)D is <10 ng/ml [severely deficient (vitamin D Council 2019)] of any 'control' patient, then he will be dropped out from the study (for ethical purpose) and a new COPD patient will be enrolled to fulfil the desired sample number. After that they will be cordially requested to visit again the Department of Physiology, BSMMU on '26th week' to reexamine all the study variables, and the data will be recorded as values of '26th week' (A2, B2).

During the entire study period (26 weeks), a good rapport will be kept by the researcher with every patient through taking time to time follow up over telephone and visiting patient's place with scheduled appointment to maintain a proper follow up at 2nd (at 13th week) and 3rd (at 26th week) visit of the study.

Any patient, who will fail to follow the study procedure exactly during study period, he will be dropped and a new one will be included to fulfil the desired total sample.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonologist diagnosed COPD patients

Duration of COPD: 1-10 years

Vitamin D3 deficient : Serum 25(OH)D <30 ng/ml

Age: >40years

Sex: Male

Socioeconomic status: Middle class

smoker

Exclusion Criteria:

* With acute exacerbation of:

any other pulmonary diseases like - bronchial asthma respiratory tract infection bronchiectasis pneumothorax pleural effusion tuberculosis pulmonary fibrosis pneumonectomy or pulmonary lobectomy any cardiac disease, like -

* unstable angina pectoris
* congestive heart failure
* myocardial infarction
* cardiac arrhythmia

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Effects of vitamin D3 supplementation on antioxidant enzymes level in vitamin D3 deficient COPD patients | 6 months vitamin D3 supplementation
  vitamin D3 supplementation will cause increased antioxidant enzymes level in vitamin D3 deficient COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Taskina Ali, MBBS,M.Phil, Study Director — Professor
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No